CLINICAL TRIAL: NCT01920035
Title: A Randomized, Controlled Study of the Use of Localized Endorectal Cooling Using the UroCool System During Robotic-Assisted Radical Prostatectomy (RARP) to Minimize Trauma and to Provide Earlier Return to Continence
Brief Title: Study of Endorectal Cooling During RARP to Minimize Trauma and Promote Earlier Return to Continence
Acronym: UroCool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ZOLL Circulation, Inc., USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IT 04-200
Record Dates: First submitted 2013-08-07; First posted 2013-08-09 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2014-11

CONDITIONS: Incontinence
Keywords: Incontinence post RARP; Surgery induced incontinence; Incontinence after prostatectomy; Neuropathy-induced incontinence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Local cooling/hypothermia (Experimental): These patients will have the UroCool device inserted prior to RARP to induce localized cooling/hypothermia of the pelvic region prior to and during RARP surgery.
  Interventions: Device: UroCool (Local cooling/hypothermia)
- Control Group: RARP without hypothermia (No Intervention): These patients will receive standard of care only for RARP surgery. They will not receive the UroCool investigational device.

INTERVENTIONS:
Device: UroCool (Local cooling/hypothermia) — These patients will receive the UroCool device which will be inserted just prior to RARP surgery. The UroCool device will be used to effect localized cooling/hypothermia of the pelvic region prior to and during RARP surgery. It will be removed at the end of surgery.
  Other Names: Cooling group; Hypothermia group; Treatment Arm; UroCool group
  Arms: Local cooling/hypothermia

SUMMARY:
Localized cooling/hypothermia using the UroCool System during robotic-assisted radical prostatectomy (RARP) surgery results in an improved overall return to continence, (defined as not wearing any protective urinary pads), compared with standard of care in men presenting for RARP.

DETAILED DESCRIPTION:
This study will assess the use of an endorectal cooling device, UroCool, to achieve controlled, local hypothermia of the pelvis. The study will evaluate the safety and effectiveness of the device in inducing hypothermia of the neuromuscular tissues impacting continence during RARP.

The UroCool system is designed to apply targeted temperature control to the pelvic anatomy during RARP. The pelvis is cooled transrectally via a closed cycle recirculation of chilled sterile saline using a single-use disposable balloon catheter connected via a circulation IV set to a control console that is covered by a current 510(k) and commercially available.

The UroCool polymeric catheter is designed to be inserted within the rectal cavity adjacent to the prostate prior to surgery and removed upon completion of surgery. It is used in conjunction with the InnerCool Console which circulates cold saline in a closed loop within the UroCool catheter to allow for therapeutic localized cooling of the prostate gland and surrounding areas during prostate surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male and a candidate for robotic assisted radical prostatectomy (RARP) for the treatment of prostate cancer
* Patient is over eighteen (>18) years of age
* Patient reads, understands and speaks English fluently (U.S. Sites only)
* Subject understands and agrees to all pre-operative preparation procedures including a "self-administered" fleet enema
* Subject understands study procedures, risks of such procedures and is willing to comply with all study procedures
* Patient is willing and able to comply with all post-surgical milestones including completing and returning post-surgery follow up questionnaires at specified intervals over a 12 month period
* Subject agrees to participate in the study and is willing to sign the written informed consent per the enrolling site's institutional procedure

Exclusion Criteria:

* Presents with baseline or has a history of urinary incontinence
* Rectal or GI pathology deemed unsuitable for placement of the treatment device by the examining physician
* Prior extensive pelvic surgery such as low anterior resection, abdominoperineal resection, or proctocolectomy continent stool pouch, or any other extensive abdominopelvic surgery that would render the patient a high-risk for complications as deemed by the surgeon
* History of prior treatment of any kind for prostate cancer; e.g. radiation therapy, cryotherapy, high-intensity focused ultrasound (HIFU), hormonal or chemotherapy
* Prior intra-operative injuries (for example: rectal injury)
* Inadequate hemostasis
* Serious concurrent medical condition likely to result in death during the next 12 months. Any other acute or chronic condition which the Investigator believes will unacceptably increase the risk of study participation or interfere with study procedures and assessments.
* Active or recent (within 1 month prior to study enrollment) participation in another investigational clinical research study or planned to be enrolled in another study of prostate therapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Improved return of overall continence. | 90 days post RARP
  The primary objective of the study is an improved return of overall continence measured at 90 days post RARP surgery. A favorable outcome would be improved overall continence in the RARP with hypothermia group versus the RARP without hypothermia group.

SECONDARY OUTCOMES:
Faster return to continence. | 30, 60 and 90 days
  The secondary objective of the study is to see if men will achieve a return to continence faster if treated with hypothermia. This will be assessed at 30, 60 and 90 days. A favorable outcome would be a reduced time to continence in the RARP with hypothermia group versus the RARP without hypothermia group.

OTHER OUTCOMES:
Reduction of overall severe incontinence | 90 days, 6 months and 12 months
  The third objective is to assess reduction of overall severe incontinence. Severe incontinence is defined as the need for 3 or more pads in a 24 hour period. This will be assessed at 90 days, 6 and 12 months. A favorable outcome would be a reduction of overall severe incontinence in the RARP with hypothermia group versus the RARP without hypothermia group.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ahlering, MD, Principal Investigator — UC Irvine; Anthony M Mullin, MD, MDDR, Study Director — Philips Healthcare/InnerCool BU
Locations (3):
- United States (2):
  - City Of Hope, Duarte, California
  - Swedish Medical Center, Seattle, Washington
- St. Antonius-Hospital Gronau GmbH, Gronau, Germany

REFERENCES:
- [Background] Liss MA, Skarecky D, Morales B, Ahlering TE. The application of regional hypothermia using transrectal cooling during radical prostatectomy: mitigation of surgical inflammatory damage to preserve continence. J Endourol. 2012 Dec;26(12):1553-7. doi: 10.1089/end.2012.0345. Epub 2012 Nov 15. PMID 23153199
- [Background] Finley DS, Chang A, Morales B, Osann K, Skarecky D, Ahlering T. Impact of regional hypothermia on urinary continence and potency after robot-assisted radical prostatectomy. J Endourol. 2010 Jul;24(7):1111-6. doi: 10.1089/end.2010.0122. PMID 20624082
- [Derived] Huynh LM, Skarecky D, Porter J, Wagner C, Witt J, Wilson T, Lau C, Ahlering TE. A Randomized Control Trial Of Anti-Inflammatory Regional Hypothermia On Urinary Continence During Robot-Assisted Radical Prostatectomy. Sci Rep. 2018 Nov 5;8(1):16352. doi: 10.1038/s41598-018-34657-4. PMID 30397236